CLINICAL TRIAL: NCT01041534
Title: Data Investigation of Bariatric Surgery and Economic Savings: Adjustable Gastric Band (AGB) Survey Study
Brief Title: Adjustable Gastric Band Survey Study
Acronym: AGB
Status: Withdrawn | Type: Observational
Why Stopped: This study did not enroll any participants
Sponsor: University of Washington (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Flum, Professor, Surgery, University of Washington
Other Study IDs: 36720; BA-08-01/Log 2 (Other: Ventura Healthcare systems, LLC); FA7014-08-2-0002 (Other Grant/Funding Number: Department of Defense, Air Force District Washington)
Record Dates: First submitted 2009-12-29; First posted 2009-12-31 (Estimated); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Morbid Obesity
Keywords: Adjustable gastric band, morbid obesity, bariatric surgery
MeSH Terms: conditions — Obesity, Morbid | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adjustable Gastric Band (AGB) surgery: Patients who have undergone adjustable gastric band (AGB) surgery at the UWMC or other sites that have agreed to cooperate with our site (letter of cooperation and HIPAA waiver approved by our IRB) between April 1, 2007 and July 1, 2008.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Two surveys are sent to patients: Adjustable gastric band (AGB) Health Survey and a quality of life survey (EQ5D)

SUMMARY:
Our aim is to complete a survey study of patients who have undergone Adjustable Gastric Band (AGB) surgery at the University of Washington Medical Center (UWMC) and expanded to other bariatric surgical sites outside the University of Washington (UW), which will obtain a HIPAA waiver and a letter of cooperation) between April 1, 2007 and July 1, 2008. (Please note the University of Washington team will not have access to the site's list of patients, only access to coded returned surveys sent back from patients). Patients will be identified by obtaining operative case lists from the Department of Surgery Quality Improvement Team who maintain monthly records of bariatric procedures performed. We will obtain patient contact information (address) and patients will be contacted by mail with the request that they complete both the Adjustable Gastric Band (AGB) Health Survey and a standard Quality of Life survey (EQ5D). The mailing will include an Information Statement, the AGB Survey, the EQ5D, and a stamped return envelope. As an incentive, a $2 bill will be sent along with the first mailing to cover the costs of completing and returning the surveys. Patients who do not return survey within 30 days will be mailed a second survey. Patients who do not return the second survey within 30 days will be mailed a third survey. Patients who do not return the third survey will not be re-contacted.

DETAILED DESCRIPTION:
While there has been considerable energy focused on the costs and effectiveness of bariatric surgery, there has been little systematically-gathered evidence on the non-surgical care and healthcare expenditures for similarly burdened patients. The economic burden and clinical impact of both need to be more carefully defined to help guide DOD decision making regarding obesity care. Understanding the cost effectiveness of obesity treatments is also critical given the cost of treatment procedures, their potential for saving future costs related to co-morbid health conditions and worker productivity and the growing population of operative candidates.

This study will provide a comprehensive assessment of the burden and costs of operative and non-operative obesity care across all regions in the U.S. where the Department of Defense (DOD) authorizes care. The development of economic assessment tools will allow health policy experts, purchasers and payers of healthcare, clinicians and patients to determine the utility and cost-effectiveness of available treatment strategies. These economic considerations are relevant to the competing crises of spiraling health care costs and the loss of productivity related to obesity.

The specific purpose of this study is to provide a comprehensive assessment of the burden and costs of operative and non-operative obesity care to develop a set of economic assessment tools that will allow health policy experts, purchasers and payers of healthcare, clinicians and patients to determine the utility and cost-effectiveness of available treatment strategies for managing obesity. Utility refers to qualitative components affected by clinical conditions such as individual's perceptions of quality of life, ability to take care of one-self, or ability to work/be productive. We anticipate that utility changes greatly for people who are able to achieve weight loss, but the differences or degree to which operative and non-operative weight loss treatments affects utility is not well known.

In particular, less is known about the effect of Adjustable Gastric Band (AGB) surgery on utility because it has only emerged as a predominant form of surgical treatment in the United States approximately within the last five years - for example, the first AGB surgery at UWMC was only performed in April 2007. In addition, assessment of cost-effectiveness of treatments requires understanding healthcare use after treatment (i.e. how many follow-up visits do you have with a doctor because of your surgical treatment) and AGB requires frequent follow-up visits in the first three years to make the surgical treatment effective. There is little information or research reporting the actual frequency of which patients are receiving follow-up care after AGB surgery, the cost for that care (is it a patient cost or insurance covered), or whether frequency of follow-up care affects long-term weight loss or health outcomes.

While the original procedures of our related study (IRB #35310, Committee E/A) only included secondary analysis of existing datasets, we have found very little information about qualitative utility or use/frequency of follow-up care for AGB patients and feel these are important aspects for modeling treatment choices for patients considering AGB. By adding a survey component, we will capture these data elements that are otherwise not found in literature or administrative datasets.

ELIGIBILITY:
Inclusion Criteria:

* All patients that have undergone Adjustable gastric band (AGB bariatric surgery) and those with diagnoses of morbid obesity will be included. All patients having a AGB bariatric operation between April 1, 2007 and July 1, 2008 will be included in this analysis except for those with exclusionary diagnoses.

Exclusion Criteria:

* Current "Longitudinal Assessment of Bariatric Surgery (LABS)" study participation (note: LABS study captures similar information on utility and frequency of healthcare use, but has not yet published data that we could otherwise incorporate into our study. All LABS study sites, as University of Washington Medical Center (UWMC) is, are prohibited from duplicating research efforts in LABS enrolled patients to reduce burden on patients and conflict of interest in research reporting)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone adjustable gastric band (AGB) surgery between April 1, 2007 and July 1, 2008 at University of Washington Medical Center (UWMC) or other sites that have been approved by our IRB (all within the Washington State area).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Flum, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States